CLINICAL TRIAL: NCT01739946
Title: Urinary Biomarkers For Objective Measurement Of InterStim® Response In Over Active Bladder (OAB) Patients.
Status: Completed | Type: Observational
Sponsor: Michael Chancellor, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Michael Chancellor, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2012-143
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Implanted subject: Subjects with Interstim implanted
- Controls: Subjects without Interstim implanted

SUMMARY:
The goal of this study is to compare protein markers in the urine of patients with and without overactive bladder (OAB) and InterStim®.

DETAILED DESCRIPTION:
This study will look for changes in protein markers that might reflect bladder symptoms before and after InterStim® implant.

ELIGIBILITY:
OAB subjects (n=10 Phase I and n=10 Phase II)

Inclusion Criteria:

* Female
* Age 18-75 years
* Clinical symptoms of OAB (urgency and frequency with or without urge incontinence) for at least 3 or the 6 months immediately before the first visit.
* At least 8 voids/day and an average of 1 nocturnal void over 3 consecutive days on baseline bladder diary.
* InterStim® treatment naïve or being revised with a new lead

Exclusion Criteria:

* Pelvic mass, pelvic prolapse, urinary retention, and pelvic malignancies as revealed by physical examination/medical record review
* Implanted Programmable Generator (IPG) is not implanted/connected to the tined lead (failed Stage I)
* Revision of only the IPG (without replacement of the tined lead)
* More than one InterStim® device being placed (undergoing bilateral stimulation)

Controls (n=10)

Inclusion:

* Female
* Age 18-75 years
* Deny history of OAB diagnosis or symptoms (urgency and frequency with or without urge incontinence)
* American Urological Association (AUA) symptom score of ≤4

Exclusion:

-History of pelvic mass, prolapse, urinary retention, or pelvic malignancy within the last year

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with either have OAB and will be undergoing an InterStim® implant (InterStim® group) or do not have bladder symptoms or an InterStim® device (Control group)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Nerve Growth Factor (NGF) levels | 4 weeks
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chancellor, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Peters KM, Jayabalan N, Bui D, Killinger K, Chancellor M, Tyagi P. Effect of Sacral Neuromodulation on Outcome Measures and Urine Chemokines in Interstitial Cystitis/Painful Bladder Syndrome Patients. Low Urin Tract Symptoms. 2015 May;7(2):77-83. doi: 10.1111/luts.12054. Epub 2014 Mar 17. PMID 26663686